CLINICAL TRIAL: NCT02577640
Title: Dietary Soy Isoflavones In Chronic Pancreatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Philip Hart, Assistant Professor-Clinical, Ohio State University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014H0226
Record Dates: First submitted 2015-10-07; First posted 2015-10-16 (Estimated); Results first posted 2021-11-12 (Actual); Last update posted 2021-11-12 (Actual); Status verified 2021-10

CONDITIONS: Chronic Pancreatitis
MeSH Terms: conditions — Pancreatitis, Chronic | interventions — Soybean Proteins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dose Escalation (DE) Phase (Experimental): Here a traditional 3+3 design will be used to determine the compliance, tolerability and dose limiting toxicities in this unique patient population. Dose escalation with soy bread will be continued until dose-limiting toxicities are observed in >33% of the participants or the daily target dose of 4 slices of bread [132 mg soy isoflavone] is reached.
  Interventions: Dietary Supplement: Soy bread
- Maximum Tolerated Dose (MTD) Phase (Experimental): After the Phase I study has been completed, an additional 10 chronic pancreatitis patients will be treated at the best tolerated dose of soy bread for 4 weeks to further verify safety and toxicity.
  Interventions: Dietary Supplement: Soy bread

INTERVENTIONS:
Dietary Supplement: Soy bread — Soy breads will be produced using a sponge-dough process. Finished dough will be formed, panned, and proofed in proofing cabinet (~95% RH) at 40ºC for 60 minutes. Proofed loaves will be baked for 50 minutes at 150ºC in a convection oven (jet air oven, model: JA14, Doyon, Liniere, Quebec, Canada). Breads will be considered done at an internal temperature of 95 ± 5ºC.
  Other Names: Soy Isoflavones

SUMMARY:
Dietary Soy Isoflavones in Chronic Pancreatitis: Investigating the Anti-inflammatory Effects of Food Innovation Science on Gastrointestinal Disease

DETAILED DESCRIPTION:
Management of pancreatic disorders imparts a major burden on healthcare costs, estimated at over 3 billion dollars annually. Chronic pancreatitis is characterized by chronic inflammation and progressive scarring, leading to abdominal pain, irreversible damage to the pancreas and the loss of both exocrine and endocrine function. Additionally, chronic pancreatic inflammation is a risk factor for pancreas cancer. There are no current treatments to modify the natural history of this disorder. Thus, identifying novel therapeutic options for this disease represents a high priority, and could fill an unmet medical need to improve quality of life, reduce risk of malignant transformation, and limit exorbitant medical costs associated with patient care. The investigators have assembled a multi-disciplinary research team to pursue an alternative, non-pharmacologic approach to limiting inflammatory cascades in (Chronic Pancreatitis) CP patients. They will assess compliance, toxicity and measure the changes in pro-inflammatory cytokine expression from a soy based dietary bread product using a classic 3+3 dose escalation study design in subjects with chronic pancreatitis.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of chronic pancreatitis by fulfilling one of the following clinical scenarios:

   1. Presence of pancreatic calcifications
   2. Suggestive for chronic pancreatitis - consistent EUS criteria or at least 3 abnormal side branches on pancreatic duct imaging
   3. Indeterminate EUS findings for chronic pancreatitis with evidence of exocrine pancreatic insufficiency (EPI)
2. Age ≥18 years

Exclusion Criteria:

1. Inability to provide written consent
2. Inability to comply with the study protocol
3. Soy allergy
4. Pancreatic cancer
5. History of prior pancreatic surgery (this does not include endoscopic therapies)
6. Comorbid diseases characterized by a chronic inflammatory state, including, but not limited to rheumatologic diseases, chronic kidney disease, extra-pancreatic malignancy
7. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-07; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip Hart, MD, Principal Investigator — The Ohio State Wexner Medical Center
Locations (1):
- Philip Hart, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ahn-Jarvis J, Lombardo E, Cruz-Monserrate Z, Badi N, Crowe O, Kaul S, Komar H, Krishna SG, Lesinski GB, Mace TA, Ramsey ML, Roberts K, Stinehart K, Traczek M, Conwell DL, Vodovotz Y, Hart PA. Reduction of inflammation in chronic pancreatitis using a soy bread intervention: A feasibility study. Pancreatology. 2020 Jul;20(5):852-859. doi: 10.1016/j.pan.2020.04.018. Epub 2020 Jun 6. PMID 32595109

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Escalation Group 1: DE group at 1 slice of bread per day.
- Dose Escalation Group 2: DE group at 2 slices of bread per day
- Dose Escalation Group 3: DE group at 3 slices of bread per day
- Maximally Tolerated Dose: maximally tolerated dose of bread for 4 week period
Period: Dose Escalation Group 1
Arm/Group | Dose Escalation Group 1 | Dose Escalation Group 2 | Dose Escalation Group 3 | Maximally Tolerated Dose
Started | 4 | 0 | 0 | 0
Completed | 3 | 0 | 0 | 0
Not Completed | 1 | 0 | 0 | 0
Period: Dose Escalation Group 2
Arm/Group | Dose Escalation Group 1 | Dose Escalation Group 2 | Dose Escalation Group 3 | Maximally Tolerated Dose
Started | 0 | 3 | 0 | 0
Completed | 0 | 3 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Dose Escalation Group 3
Arm/Group | Dose Escalation Group 1 | Dose Escalation Group 2 | Dose Escalation Group 3 | Maximally Tolerated Dose
Started | 0 | 0 | 3 | 0
Completed | 0 | 0 | 3 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Maximally Tolerated Dose
Arm/Group | Dose Escalation Group 1 | Dose Escalation Group 2 | Dose Escalation Group 3 | Maximally Tolerated Dose
Started | 0 | 0 | 0 | 1
Completed | 0 | 0 | 0 | 1
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: A total of 8 unique subjects were enrolled into the DE phase. One subject was a screen failure due to pre-existing solid food dysphagia, which was not reported at screening. For each of the three doses, three subjects completed all study activities; two subjects completed both dose escalation group 1 and 3.
  One additional unique subject completed the MTD phases consuming 3 slices per day for 4 weeks.
Groups:
- Dose Escalation Group 1: 1 slice bread per day for 1 week
- Dose Escalation Group 2: 2 slices bread per day for 1 week
- Dose Escalation Group 3: 3 slices bread per day for 1 week
- Maximally Tolerated Dose: maximally tolerated dose for 4 weeks
- Total: Total of all reporting groups
Arm/Group | Dose Escalation Group 1 | Dose Escalation Group 2 | Dose Escalation Group 3 | Maximally Tolerated Dose | Total
Number analyzed (Participants) | 4 | 3 | 1 | 1 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 0 | 1 | 0 | 3
  >=65 years | 2 | 3 | 0 | 1 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 0 | 0 | 2
  Male | 3 | 2 | 1 | 1 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 0 | 0 | 3
  White | 2 | 2 | 1 | 1 | 6
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Dose Limiting Toxicities
Description: Participants were evaluated for the development of bothersome symptoms that prevented them from being able to complete the recommended intervention course. Counts represent number of subjects who developed a symptom that prevented the ability to complete the dose/study period.
Time Frame: 1 (dose escalation groups) or 4 (maximally tolerated dose) weeks
Measure: Count of Participants; unit: Participants
Groups:
- Dose Escalation Group 1: 1 slice bread per day
- Dose Escalation Group 2: 2 slices per day
- Dose Escalation Group 3: 3 slices per day
- Maximally Tolerated Dose Group: maximally tolerated dose (3 slices/day)
Arm/Group | Dose Escalation Group 1 | Dose Escalation Group 2 | Dose Escalation Group 3 | Maximally Tolerated Dose Group
Number analyzed (Participants) | 3 | 3 | 3 | 1
Participants | 0 | 0 | 0 | 0

2. Secondary Outcome: Pro-inflammatory Cytokines
Description: Changes in the serum were assessed for TNF-alpha prior to and following introduction of soy bread
Time Frame: 1 (dose escalation group) or 4 weeks (maximally tolerated subject)
Population: For the purposes of analyzing the secondary outcomes all subjects completing any of the dose escalation groups were combined.
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- Dose Escalation (DE) Phase: Data for each of the 3 doses were examined collectively.
- Maximum Tolerated Dose (MTD) Phase: Actual data for subjects who completed MTD phase over 4 weeks.
Arm/Group | Dose Escalation (DE) Phase | Maximum Tolerated Dose (MTD) Phase
Number analyzed (Participants) | 9 | 1
pg/mL
  Day 0 value of TNF-alpha | 2.67 (0.72) | 7.0 (0)
  Day 7 value of TNF-alpha | 2.38 (0.56) | 7.2 (0)

ADVERSE EVENTS:
Time Frame: up to 4 weeks
Groups:
- Dose Escalation Group 1: 1 slice per day
- Maximally Tolerated Dose: an extended exposure to the maximally tolerated dose of 3 slices per day.
Arm/Group | Dose Escalation Group 1 | Dose Escalation Group 2 | Dose Escalation Group 3 | Maximally Tolerated Dose
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/1
Other Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-12-05): https://cdn.clinicaltrials.gov/large-docs/40/NCT02577640/Prot_SAP_000.pdf